CLINICAL TRIAL: NCT07135089
Title: Improving Neuroprotective Strategy for Ischemic Stroke Before Endovascular Thrombectomy by Intravenous Tirofiban (INSIST-IT2): a Prospective, Randomized, Double Blinded, Multi-center Study
Brief Title: Improving Neuroprotective Strategy for Ischemic Stroke Before Endovascular Thrombectomy by Intravenous Tirofiban
Acronym: INSIST-IT2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Y(2025)114
Record Dates: First submitted 2025-08-12; First posted 2025-08-21 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): Intravenous tirofiban before endovascular thrombectomy
  Interventions: Drug: Intravenous tirofiban before endovascular thrombectomy
- Placebo group (Placebo Comparator): Intravenous placebo before Endovascular Thrombectomy
  Interventions: Drug: Intravenous placebo before endovascular thrombectomy

INTERVENTIONS:
Drug: Intravenous tirofiban before endovascular thrombectomy — The tirofiban was administrated as a bolus dose of 10 μg/kg, followed by continuous infusion of 0.15 μg/kg/min for up to 24 hours.
  Arms: Tirofiban group
Drug: Intravenous placebo before endovascular thrombectomy — The placebo was administrated as a bolus dose of 10 μg/kg, followed by continuous infusion of 0.15 μg/kg/min for up to 24 hours.
  Arms: Placebo group

SUMMARY:
It remains uncertain whether intravenous tirofiban administered before endovascular thrombectomy could improve disability severity for patients with LVO due to intracranial atherosclerosis.The current study aimed to assess the efficacy and safety of administering intravenous tirofiban before endovascular thrombectomy for improving clinical outcomes in patients with anterior circulation LVO due to intracranial atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Anterior circulation large vessel occlusion (the internal carotid artery or the first or second segment of the middle cerebral artery) confirmed by computed tomography angiography (CTA) or magnetic resonance angiography (MRA);
* Eligible for endovascular treatment within 12 hours of symptom onset;
* Based on the patient's medical history, clinical presentation, and imaging findings, large artery atherosclerosis is highly suspected as the underlying etiology;
* Baseline National Institute of Health Stroke Scale (NIHSS) ≥ 6;
* Baseline ASPECTS ≥ 6 on CT;
* A pre-stroke modified Rankin Scale (mRS) score of ≤2;
* Signed informed consent by patient or their legally authorized representative.

Exclusion Criteria:

* History of atrial fibrillation or atrial flutter, or 12-lead Electrocardiogram before randomization and after admission showing atrial flutter or atrial fibrillation;
* Hemorrhagic stroke: cerebral hemorrhage, subarachnoid hemorrhage, or a history of bleeding within one month;
* Intracranial aneurysms or malformations, tortuous arteries that hinder thrombectomy, and space-occupying effect brain tumors;
* The following drugs are taken within one week: dual antiplatelet drugs, direct oral anticoagulants (DOACs), warfarin and other drugs that increase the risk of bleeding;
* Severe uncontrolled hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg);
* Deficiency of anticoagulant factors or international normalized ratio (INR) > 1.7, platelet count < 90×10⁹/L;;
* Severe renal insufficiency and advanced disease with an expected life expectancy of less than 6 months;
* Pregnancy or lactation;
* Allergy to drugs or contrast agents;
* Participating in other clinical trials;
* Other conditions that the researcher deems unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with functional independence (modified Rankin Scale [mRS] score of 0 to 2) | Day 90
  mRS ranges from 0-6, with high score meaning poor outcome

SECONDARY OUTCOMES:
The proportion of patients without disability (modified Rankin Scale [mRS] score of 0 to 1) or who returned to their premorbid mRS score at 90 days (for patients with prestroke mRS score >1) | Day 90
  mRS ranges from 0-6, with high score meaning poor outcome
ordinal distribution of modified Rankin Scale (mRS) | Day 90
  mRS ranges from 0-6, with high score meaning poor outcome
The proportions of patients with substantial reperfusion at initial preprocedure catheter angiogram (defined as mTICI score ≥2b) | immediately after first catheter angiogram
  Substantial reperfusion was defined as an expanded Thrombolysis In Cerebral Infarction grade of 2b50 (substantial reperfusion), 2c (nearcomplete reperfusion), or 3 (complete reperfusion).
The proportions of patients with substantial reperfusion at final angiogram | immediately after final angiogram
The proportions of patients with complete recanalization as assessed by CTA or MRA 48 hours after endovascular treatment | 24 (-6/+24) hours
Change in National Institute of Health stroke scale (NIHSS) | 24 (-6/+24) hours
  NIHSS ranges from 0-42, with high score meaning poor outcome
change in National Institute of Health stroke scale (NIHSS) | 7 (-2/+2) days
  NIHSS ranges from 0-42, with high score meaning poor outcome
The incidence of symptomatic intracranial hemorrhage assessed according to Heidelberg bleeding classification | 24 (-6/+24) hours
The incidence of intraparenchymal hemorrhage (PH1 and PH2) | 24 (-6/+24) hours
The incidence of non-intracranial hemorrhage complications | 24 (-6/+24) hours
Serious adverse events | 7 (-2/+2) days
  eg, acute respiratory failure, large or malignant middle cerebral artery infarction, acute heart failure, hemicraniectomy
Procedure-associated complications | Periprocedural
The proportion of patients with thrombocytopenia | 24 (-6/+24) hours
The incidence of mortality | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided